CLINICAL TRIAL: NCT00120809
Title: A Randomised, Placebo Controlled Trial of Intermittent Preventative Treatment With Sulfadoxine-pyrimethamine in Gambian Multigravidae.
Brief Title: Intermittent Preventative Treatment With Sulfadoxine-Pyrimethamine in Gambian Multigravidae
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Department of State for Health and Social Welfare, The Gambia (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ITCRVG27b
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Multigravidae; Intermittent preventative treatment; Sulfadoxine-pyrimethamine
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine

SUMMARY:
Malaria is particularly harmful during pregnancy causing anemia in the mother and low birth weight which, in turn, increases infant mortality. Thus, the World Health Organization (WHO) now recommends that all pregnant women who live in malaria endemic areas of Africa should receive sulfadoxine-pyrimethamine (SP) at monthly intervals during the second and third trimesters of pregnancy. Malaria is especially severe during first pregnancies and the value of intermittent preventative treatment with SP during first pregnancies has been clearly shown. However, it is less certain whether multigravidae, who are at less risk, also benefit from intermittent preventative treatment with SP. To investigate this, a trial has been conducted in Gambian multigravidae who were given intermittent preventative treatment with SP or placebo during the second and third trimesters. The prevalence of anemia six weeks after delivery, low birth weight and poor outcome of pregnancy in women in each group were studied.

DETAILED DESCRIPTION:
Objective

The objective of this study was to determine whether intermittent preventative treatment (IPTp) with sulfadoxine-pyrimethamine (SP) reduced the prevalence of anemia and low birth weight in Gambian multigravidae.

Study area

The study was carried out in 14 mother and child health (MCH) clinics situated on the north and south banks of the River Gambia near to the town of Farafenni in the centre of the country. In this area, malaria is highly seasonal with an entomological inoculation rate of 10 -50 infectious bites per year.

Study population

All women who attended one of the study clinics during the trial period and who were multigravidae were asked if they wished to join the study. If this was the case, an initial screening questionnaire was administered to assess their suitability to do so. Eligibility criteria were - a pregnancy of more than 15 weeks gestation, a hemoglobin (Hb) concentration of more than 7 g/dL, absence of a history of sensitivity to sulfonamides and absence of any chronic underlying illness.

Randomisation

If a woman met the eligibility criteria, informed written consent was sought and, if this was given, the woman was formally recruited to the study and allocated a trial number and randomised to receive either SP or placebo. Randomisation was done in blocks of 12; each field worker was assigned a number of blocks to ensure balanced recruitment between centers.

Drug administration

Women were allocated to receive SP (pyrimethamine 25 mg + sulfadoxine 500 mg)(Cosmos Pharmaceuticals, Nairobi) or matching placebo. An initial dose of SP or placebo (three tablets) was given at the time of enrolment into the trial and at all subsequent visits to the antenatal clinic up to a maximum of four treatments. All women were given iron and folic acid supplements as recommended by the Ministry of Health guidelines.

Surveillance

Women were visited at home twice per week by a project field worker to assess their health and to encourage them to attend the ante-natal clinic at monthly intervals. Women with a high risk of obstetric complications were encouraged to deliver in hospital but most women delivered at home.

If a delivery occurred in hospital or a health center a finger prick blood sample was obtained and the birth weight was measured. In the case of women who delivered at home, the weight of the new born baby was measured within 5 days of delivery and a finger prick blood sample obtained for measurement of Hb concentration and preparation of blood films.

Women were visited at home six weeks after delivery when an additional blood sample was obtained and one year later to investigate the health of their child.

Laboratory methods

Hemoglobin concentration was measured using a Hemocue (Hemocue AB, Angelholm, Sweden). Thick blood films were stained with Giemsa and examined for malaria parasites. Each slide was read by two microscopists. If discrepant results were obtained, the slide was read by a third microscopist and the majority view accepted.

Trial end-points

The co-primary trial end-points were hemoglobin concentration at, or shortly after, birth and birthweight or weight of the baby shortly after birth.

Sample size

To detect a 20% reduction in the estimated risk of severe anemia (Hb <7 g/dl) among multigravidae, estimated to be 30% in the control group, with 80 % power at the 5% level of significance and allowing for a 30% loss to follow-up it was calculated that a study with 1115 women in each arm was required. To show a reduction in the proportion of low birthweight babies from the expected 18% in the control group to 12% in the SP group with 80% power it was estimated that 2 x 1538 women would be needed. Thus, the target sample size was 3,000.

Data management and analysis

All data were double entered and verified. Prior to the breaking of the code the data base was locked and a copy given to the chair of the Data Safety Monitoring Board (DSMB). Statistical analysis was done using S-plus and STATA. An analytical plan was prepared and approved by the DSMB before the code was broken.

Trial oversight

The trial was monitored by a DSMB. It was conducted in line with the requirements of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Multigravid pregnancy.
* Residence in study area.
* Informed consent.

Exclusion Criteria:

* Allergy to sulfonamides.
* Chronic illness.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000
Dates: Start 2002-07; Study Completion 2004-09

PRIMARY OUTCOMES:
Hemoglobin concentration at delivery.
Birthweight.

SECONDARY OUTCOMES:
Hemoglobin concentration six weeks after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Greenwood, MD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- Medical Research Council Laboratories, Banjul, The Gambia